CLINICAL TRIAL: NCT00463333
Title: Postoperative Delirium at Heidelberg's Intensive Care Unit -New Diagnostic Markers
Status: Completed | Type: Observational
Sponsor: Heidelberg University (Other)
Collaborators: Else Kröner Fresenius Foundation (Other)
Other Study IDs: 196/2004
Record Dates: First submitted 2005-09-10; First posted 2007-04-20 (Estimated); Last update posted 2007-04-20 (Estimated); Status verified 2007-04

CONDITIONS: Postoperative Delirium
Keywords: postoperative delirium; psychometric testing; EEG; serum markers
MeSH Terms: conditions — Emergence Delirium

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Summary:

Postoperative delirium is a highly prevalent disease (10-30% prevalence) after surgery in intensive care unit, however, it is often misdiagnosed and mistreated. The aim of the present project is to investigate risk factors for postoperative delirium in more detail, to evaluate respective cognitive test systems and to measure EEG activity parallel to patients' serum anticholinergic activity. The pathophysiology of delirium is unknown up to now: a possible dysbalance between cerebral acetylcholine and dopamine concentrations is a likely hypothesis. Therefore, the measurement of peripheral serum anticholinergic activity could be a new prognostic factor for evaluation of delirium. Because delirium is also associated with higher postoperative mortality and morbidity, with delayed functional recovery, and postoperative delirium makes patient management much more difficult, increases costs, and, above all, causes severe discomfort to the patient new interdisciplinary diagnostic strategies are necessary to resolve this problem.

ELIGIBILITY:
Inclusion Criteria:

* All patients at Intensive Care Unit over a defined time period
* Over 18 years old

Exclusion Criteria:

* Elective heart and vascular patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2005-05

CONTACTS AND LOCATIONS:
Overall Officials: Markus A Weigand, PhD, MD, Principal Investigator — Medical Faculty, Clinic of Anesthesiology, University of Heidelberg; Konstanze Plaschke, Prof., Principal Investigator — Clinic of Anesthesiology
Locations (1):
- Intensive Care Unit, Clinic of Anesthesiology, Heidelberg, Heidelberg, Germany

REFERENCES:
- [Derived] Plaschke K, Kopitz J, Mattern J, Martin E, Teschendorf P. Increased cortisol levels and anticholinergic activity in cognitively unimpaired patients. J Neuropsychiatry Clin Neurosci. 2010 Fall;22(4):433-41. doi: 10.1176/jnp.2010.22.4.433. PMID 21037129